CLINICAL TRIAL: NCT01936181
Title: A Randomised, Double-blind, Parallel Group, Multicentre Clinical Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Immunogenicity of SB2 Compared to Remicade® in Subjects With Moderate to Severe Rheumatoid Arthritis Despite Methotrexate Therapy
Brief Title: A Study Comparing SB2 to Remicade® in Subjects With Moderate to Severe Rheumatoid Arthritis Despite Methotrexate Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB2-G31-RA
Record Dates: First submitted 2013-09-02; First posted 2013-09-05 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Infliximab; Biosimilar
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SB2 (proposed biosimilar to inflixmab) (Experimental): SB2 3 mg/kg at week 0, 2, 6 then every 8 weeks thereafter via intravenous infusion up to Week 70
  Interventions: Drug: SB2 (proposed biosimilar to infliximab)
- Remicade (infliximab) (Active Comparator): Remicade 3 mg/kg at week 0, 2, 6 then every 8 weeks thereafter via intravenous infusion up to Week 46
  Interventions: Drug: Remicade (infliximab)
- Remicade (infliximab), switch to SB2 (Experimental): SB2 3mg/kg at week 54, 62, 70
  Interventions: Drug: SB2 (proposed biosimilar to infliximab)
- Remicade (infliximab), continue as Remicade (Active Comparator): Remicade 3mg/kg at week 54, 62, 70
  Interventions: Drug: Remicade (infliximab)

INTERVENTIONS:
Drug: Remicade (infliximab)
  Arms: Remicade (infliximab); Remicade (infliximab), continue as Remicade
Drug: SB2 (proposed biosimilar to infliximab)
  Arms: Remicade (infliximab), switch to SB2; SB2 (proposed biosimilar to inflixmab)

SUMMARY:
This is a randomized, double-blind, parallel group, multicentre clinical study to evaluate the efficacy, safety, pharmacokinetics and immunogenicity of SB2 compared to Remicade in subjects with moderate to severe Rheumatoid Arthritis (RA) despite Methotrexate (MTX) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as having RA according to the revised 1987 ACR criteria for at least 6 months
* Have moderate to severe active disease despite MTX therapy defined as having more than or equal to six swollen joints and more than or equal to six tender joints and either erythrocyte sedimentation rate (ESR, Westergren) ≥ 28 mm/h or serum C-reactive protein ≥ 1.0 mg/dL
* Must have been treated with MTX for at least 6 months prior to Randomisation and on a stable dose of MTX 10-25 mg/week given at least 4 weeks prior to Screening
* Female subjects who are not pregnant or nursing at Screening and who are not planning to become pregnant from Screening until 6 months after the last dose of investigational product

Inclusion Criteria for Transition-Extension Period:

* Have been enrolled and completed the scheduled Week 54 visit of the randomised, double-blind period of the SB2-G31-RA study
* In the opinion of the Investigator, subjects who may benefit from continuing IP treatment (either SB2 or Remicade), understand the implications of taking part in the study and willing to participate in the transition-extension period

Exclusion Criteria:

* Have been treated previously with any biological agents including any tumour necrosis factor inhibitor
* Have a known hypersensitivity to human immunoglobulin proteins or other components of Remicade or SB2
* Have a positive serological test for hepatitis B or hepatitis C or have a known history of infection with human immunodeficiency virus
* Have a current diagnosis of active tuberculosis
* Have had a serious infection or have been treated with intravenous antibiotics for an infection within 8 weeks or oral antibiotics within 2 weeks prior to Randomisation.
* Have any of the following conditions

  1. Other inflammatory or rheumatic diseases.
  2. History of any malignancy within the previous 5 years prior to Screening
  3. History of lymphoproliferative disease including lymphoma.
  4. History of congestive heart failure
  5. Physical incapacitation (ACR functional Class IV or wheelchair-/bed-bound).
  6. History of demyelinating disorders.

Exclusion Criteria for Transition-Extension Period:

* Have been withdrawn from the SB2-G31-RA study for any reason
* Have had any significant medical conditions, such as an occurrence of a serious AE (SAE) or intolerance of SB2 or Remicade during the randomised, double-blind period of the SB2-G31-RA study which may render the subject unsuitable to participate in the transition-extension period, at the discretion of the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Yoon Choe, M.D., Ph.D., Principal Investigator — Daegu Catholic University Medical Center
Locations (2):
- Investigational Site, Hristo Botev Str., Sliven, Bulgaria
- Investigational Site, Santariskiu, Vilnius County, Lithuania

REFERENCES:
- [Derived] Smolen JS, Choe JY, Weinblatt ME, Emery P, Keystone E, Genovese MC, Myung G, Hong E, Baek I, Ghil J. Pooled analysis of TNF inhibitor biosimilar studies comparing radiographic progression by disease activity states in rheumatoid arthritis. RMD Open. 2020 Jan;6(1):e001096. doi: 10.1136/rmdopen-2019-001096. PMID 31958281
- [Derived] Smolen JS, Choe JY, Prodanovic N, Niebrzydowski J, Staykov I, Dokoupilova E, Baranauskaite A, Yatsyshyn R, Mekic M, Porawska W, Ciferska H, Jedrychowicz-Rosiak K, Zielinska A, Lee Y, Rho YH. Safety, immunogenicity and efficacy after switching from reference infliximab to biosimilar SB2 compared with continuing reference infliximab and SB2 in patients with rheumatoid arthritis: results of a randomised, double-blind, phase III transition study. Ann Rheum Dis. 2018 Feb;77(2):234-240. doi: 10.1136/annrheumdis-2017-211741. Epub 2017 Oct 17. PMID 29042358
- [Derived] Smolen JS, Choe JY, Prodanovic N, Niebrzydowski J, Staykov I, Dokoupilova E, Baranauskaite A, Yatsyshyn R, Mekic M, Porawska W, Ciferska H, Jedrychowicz-Rosiak K, Zielinska A, Choi J, Rho YH. Comparing biosimilar SB2 with reference infliximab after 54 weeks of a double-blind trial: clinical, structural and safety results. Rheumatology (Oxford). 2017 Oct 1;56(10):1771-1779. doi: 10.1093/rheumatology/kex254. PMID 28957563
- [Derived] Choe JY, Prodanovic N, Niebrzydowski J, Staykov I, Dokoupilova E, Baranauskaite A, Yatsyshyn R, Mekic M, Porawska W, Ciferska H, Jedrychowicz-Rosiak K, Zielinska A, Choi J, Rho YH, Smolen JS. A randomised, double-blind, phase III study comparing SB2, an infliximab biosimilar, to the infliximab reference product Remicade in patients with moderate to severe rheumatoid arthritis despite methotrexate therapy. Ann Rheum Dis. 2017 Jan;76(1):58-64. doi: 10.1136/annrheumdis-2015-207764. Epub 2015 Aug 28. PMID 26318384

RESULTS

PARTICIPANT FLOW:
Groups:
- SB2 (Proposed Biosimilar to Inflixmab): SB2 3 mg/kg at week 0, 2, 6 then every 8 weeks thereafter via intravenous infusion up to Week 70
  SB2 (proposed biosimilar to infliximab)
- Remicade (Infliximab): Remicade 3 mg/kg at week 0, 2, 6 then every 8 weeks thereafter via intravenous infusion up to Week 46
  At Week 54, subjects were randomised again in a 1:1 ratio to either continue on Remicade (Remicade/Remicade) or be transitioned to SB2 (Remicade/SB2) up to Week 70.
- Remicade (Infliximab), Switch to SB2: SB2 3mg/kg at week 54, 62, 70
  SB2 (proposed biosimilar to infliximab)
- Remicade (Infliximab), Continue as Remicade: Remicade 3mg/kg at week 54, 62, 70
  Remicade (infliximab)
Period: Randomised, Double-blind
Arm/Group | SB2 (Proposed Biosimilar to Inflixmab) | Remicade (Infliximab) | Remicade (Infliximab), Switch to SB2 | Remicade (Infliximab), Continue as Remicade
Started | 291 | 293 | 0 | 0
Completed | 227 | 225 | 0 | 0
Not Completed | 64 | 68 | 0 | 0
Not completed — Adverse Event | 27 | 21 | 0 | 0
Not completed — Protocol Violation | 1 | 5 | 0 | 0
Not completed — Lack of Efficacy | 5 | 6 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Physician Decision | 4 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 23 | 26 | 0 | 0
Not completed — Subjects from Eastern Ukraine sites | 4 | 4 | 0 | 0
Period: Transition-extension
Arm/Group | SB2 (Proposed Biosimilar to Inflixmab) | Remicade (Infliximab) | Remicade (Infliximab), Switch to SB2 | Remicade (Infliximab), Continue as Remicade
Started | 201 | 0 | 94 | 101
Completed | 186 | 0 | 88 | 96
Not Completed | 15 | 0 | 6 | 5
Not completed — Adverse Event | 3 | 0 | 3 | 1
Not completed — Lost to Follow-up | 3 | 0 | 1 | 2
Not completed — Physician Decision | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB2 (Proposed Biosimilar to Inflixmab) | Remicade (Infliximab) | Total
Number analyzed (Participants) | 291 | 293 | 584
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (11.92) | 52.6 (11.74) | 52.1 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232 | 236 | 468
  Male | 59 | 57 | 116

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology 20% Response Criteria (ACR20)
Time Frame: Week 30
Measure: Number; unit: percentage of participants
Arm/Group | SB2 (Proposed Biosimilar to Inflixmab) | Remicade (Infliximab)
Number analyzed (Participants) | 231 | 247
percentage of participants | 64.1 | 66.0

2. Secondary Outcome: ACR20
Time Frame: Week 54, Week 78
Measure: Number; unit: percentage of participants
Groups:
- SB2 at Week 54; SB2 at Week 78: SB2 3 mg/kg at week 0, 2, 6 then every 8 weeks thereafter via intravenous infusion up to Week 70
  SB2 (proposed biosimilar to infliximab)
- Remicade (Infliximab) at Week 54: Remicade 3 mg/kg at week 0, 2, 6 then every 8 weeks thereafter via intravenous infusion up to Week 46
- Remicade (Infliximab), Switch to SB2 at Week 78: Remicade 3 mg/kg at week 0, 2, 6 then every 8 weeks thereafter via intravenous infusion up to Week 46
  At Week 54, subjects were randomised to be transitioned to SB2 (Remicade/SB2) up to Week 70 and received SB2 3mg/kg at week 54, 62, 70.
  SB2 (proposed biosimilar to infliximab)
- Remicade (Infliximab), Continue as Remicade: Remicade 3 mg/kg at week 0, 2, 6 then every 8 weeks thereafter via intravenous infusion up to Week 46
  At Week 54, subjects were randomised to continue on Remicade (Remicade/Remicade) up to Week 70 and received Remicade 3mg/kg at week 54, 62, 70.
Arm/Group | SB2 at Week 54 | Remicade (Infliximab) at Week 54 | SB2 at Week 78 | Remicade (Infliximab), Switch to SB2 at Week 78 | Remicade (Infliximab), Continue as Remicade
Number analyzed (Participants) | 202 | 208 | 180 | 85 | 93
percentage of participants | 65.3 | 69.2 | 68.3 | 63.5 | 68.8

3. Secondary Outcome: American College of Rheumatology 50% Response Criteria (ACR50)
Time Frame: Week 30, Week 54, Week 78
Reporting Status: Not Posted

4. Secondary Outcome: Disease Activity Score Based on a 28 Joint Count (DAS28)
Time Frame: Week 30, Week 54, Week 78
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | SB2 (Proposed Biosimilar to Inflixmab) | Remicade (Infliximab)
All-Cause Mortality (participants affected / at risk) | 0/290 | 1/293
Serious Adverse Events (participants affected / at risk) | 36/290 | 38/293
Other Adverse Events (participants affected / at risk) | 201/290 | 203/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB2 (Proposed Biosimilar to Inflixmab) (N=290) | Remicade (Infliximab) (N=293)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Left Ventricular Failure (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus Paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Wall Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary Gland Calculus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Device Damage (General disorders) | 1 (1) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Anaphylactic Shock (Immune system disorders) | 0 (0) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pseudomembranous Colitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Soft Tissue Infection (Infections and infestations) | 1 (1) | 0 (0)
Tuberculous Pleurisy (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Arthritis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Diabetic Foot Infection (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Haematoma Infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periprosthetic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lip And/Or Oral Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar Insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian Cyst Torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB2 (Proposed Biosimilar to Inflixmab) (N=290) | Remicade (Infliximab) (N=293)
Leukopenia (Blood and lymphatic system disorders) | 4 (5) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (4)
Thrombocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anaemia Of Chronic Disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (5)
Coronary Artery Disease (Cardiac disorders) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 2 (3)
Left Ventricular Failure (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cerumen Impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Hearing Impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 3 (3) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 6 (6)
Eye Pruritus (Eye disorders) | 2 (2) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 1 (1)
Eyelid Exfoliation (Eye disorders) | 1 (1) | 0 (0)
Eyelid Oedema (Eye disorders) | 1 (1) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Lacrimation Increased (Eye disorders) | 1 (2) | 0 (0)
Myopia (Eye disorders) | 1 (1) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Presbyopia (Eye disorders) | 1 (1) | 0 (0)
Retinopathy Hypertensive (Eye disorders) | 1 (1) | 0 (0)
Visual Impairment (Eye disorders) | 1 (1) | 0 (0)
Chorioretinopathy (Eye disorders) | 0 (0) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Erythema Of Eyelid (Eye disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (4)
Abdominal Pain Upper (Gastrointestinal disorders) | 5 (7) | 6 (6)
Abdominal Pain (Gastrointestinal disorders) | 3 (4) | 3 (3)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 (3) | 4 (4)
Toothache (Gastrointestinal disorders) | 3 (4) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (3)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis Erosive (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (3) | 7 (7)
Epigastric Discomfort (Gastrointestinal disorders) | 1 (2) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastric Polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ileus Paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Submaxillary Gland Enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Wall Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis Atrophic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ileal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large Intestine Polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary Gland Calculus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 1 (1)
Chest Discomfort (General disorders) | 3 (3) | 0 (0)
Chest Pain (General disorders) | 3 (7) | 1 (1)
Chills (General disorders) | 3 (3) | 3 (5)
Oedema Peripheral (General disorders) | 3 (3) | 4 (4)
Pyrexia (General disorders) | 3 (3) | 9 (11)
Spinal Pain (General disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 2 (2)
Device Damage (General disorders) | 1 (1) | 0 (0)
Face Oedema (General disorders) | 1 (1) | 0 (0)
Influenza Like Illness (General disorders) | 1 (1) | 1 (1)
Injection Site Hypersensitivity (General disorders) | 1 (1) | 0 (0)
Injection Site Pruritus (General disorders) | 1 (1) | 0 (0)
Local Swelling (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Nodule (General disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 1 (1)
Feeling Cold (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Impaired Healing (General disorders) | 0 (0) | 1 (1)
Injection Site Rash (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary Colic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis Chronic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis Toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver Disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 3 (3) | 3 (3)
Allergy To Arthropod Sting (Immune system disorders) | 2 (2) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 2 (2) | 0 (0)
Anaphylactic Shock (Immune system disorders) | 0 (0) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Food Allergy (Immune system disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 26 (34) | 25 (34)
Latent Tuberculosis (Infections and infestations) | 24 (31) | 27 (33)
Bronchitis (Infections and infestations) | 13 (15) | 15 (18)
Upper Respiratory Tract Infection (Infections and infestations) | 13 (15) | 18 (31)
Urinary Tract Infection (Infections and infestations) | 8 (8) | 7 (7)
Pneumonia (Infections and infestations) | 7 (7) | 8 (8)
Pharyngitis (Infections and infestations) | 6 (7) | 9 (12)
Cystitis (Infections and infestations) | 3 (3) | 4 (4)
Herpes Zoster (Infections and infestations) | 3 (3) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 4 (6)
Respiratory Tract Infection (Infections and infestations) | 3 (3) | 2 (2)
Rhinitis (Infections and infestations) | 3 (3) | 5 (5)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1)
Herpes Virus Infection (Infections and infestations) | 2 (2) | 0 (0)
Oral Herpes (Infections and infestations) | 2 (3) | 3 (6)
Periodontitis (Infections and infestations) | 2 (2) | 0 (0)
Pulpitis Dental (Infections and infestations) | 2 (2) | 0 (0)
Acute Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (2) | 2 (2)
Paronychia (Infections and infestations) | 1 (1) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pseudomembranous Colitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis Chronic (Infections and infestations) | 1 (1) | 0 (0)
Schistosomiasis (Infections and infestations) | 1 (1) | 0 (0)
Soft Tissue Infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 7 (13)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0)
Tuberculous Pleurisy (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 5 (6)
Abscess Limb (Infections and infestations) | 0 (0) | 1 (1)
Arthritis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Atypical Mycobacterial Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Dacryocystitis (Infections and infestations) | 0 (0) | 1 (1)
Diabetic Foot Infection (Infections and infestations) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Haematoma Infection (Infections and infestations) | 0 (0) | 1 (1)
Lyme Disease (Infections and infestations) | 0 (0) | 2 (2)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 3 (4)
Otitis Media Acute (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Rash Pustular (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous Abscess (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Vaginal Infection (Infections and infestations) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle Rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stab Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Periprosthetic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 27 (32) | 14 (15)
Aspartate Aminotransferase Increased (Investigations) | 16 (18) | 15 (15)
Lymphocyte Count Decreased (Investigations) | 7 (8) | 2 (3)
Gamma-Glutamyltransferase Increased (Investigations) | 5 (5) | 4 (4)
Neutrophil Count Increased (Investigations) | 4 (5) | 0 (0)
Blood Creatinine Increased (Investigations) | 3 (3) | 2 (2)
Blood Pressure Increased (Investigations) | 3 (3) | 1 (1)
Blood Alkaline Phosphatase Increased (Investigations) | 2 (2) | 1 (1)
Blood Bilirubin Increased (Investigations) | 2 (2) | 1 (2)
Haemoglobin Decreased (Investigations) | 2 (2) | 1 (1)
Neutrophil Count Decreased (Investigations) | 2 (2) | 0 (0)
Transaminases Increased (Investigations) | 2 (3) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 2 (5) | 2 (4)
Aspiration Joint (Investigations) | 1 (2) | 0 (0)
Blood Calcium Increased (Investigations) | 1 (1) | 0 (0)
Blood Glucose Increased (Investigations) | 1 (1) | 4 (4)
Blood Phosphorus Decreased (Investigations) | 1 (1) | 1 (1)
C-Reactive Protein Increased (Investigations) | 1 (1) | 1 (1)
Glucose Urine (Investigations) | 1 (1) | 1 (1)
Granulocyte Count Decreased (Investigations) | 1 (1) | 0 (0)
International Normalised Ratio Decreased (Investigations) | 1 (1) | 0 (0)
International Normalised Ratio Increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte Count Increased (Investigations) | 1 (1) | 0 (0)
Platelet Count Decreased (Investigations) | 1 (1) | 0 (0)
Vitamin B12 Decreased (Investigations) | 1 (1) | 0 (0)
White Blood Cell Count Increased (Investigations) | 1 (1) | 1 (1)
Alanine Aminotransferase Abnormal (Investigations) | 0 (0) | 1 (1)
Antinuclear Antibody Increased (Investigations) | 0 (0) | 2 (2)
Antinuclear Antibody Positive (Investigations) | 0 (0) | 2 (2)
Blood Cholesterol Increased (Investigations) | 0 (0) | 1 (1)
Blood Potassium Increased (Investigations) | 0 (0) | 2 (2)
Body Temperature Increased (Investigations) | 0 (0) | 1 (1)
Double Stranded Dna Antibody (Investigations) | 0 (0) | 2 (2)
Electrocardiogram Abnormal (Investigations) | 0 (0) | 1 (1)
Haematocrit Decreased (Investigations) | 0 (0) | 1 (1)
Haematology Test Abnormal (Investigations) | 0 (0) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 2 (2)
Liver Function Test Abnormal (Investigations) | 0 (0) | 1 (1)
Red Blood Cell Count Decreased (Investigations) | 0 (0) | 1 (1)
Red Blood Cell Sedimentation Rate Increased (Investigations) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 0 (0) | 2 (3)
Weight Increased (Investigations) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 24 (30) | 15 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 9 (11)
Back Pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 14 (16)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (11)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1 (11) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Lupus-Like Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid Nodule (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Ligament Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis Postmenopausal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Eye Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal Submucosal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma Of Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign Neoplasm Of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lip And/Or Oral Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 16 (30) | 15 (16)
Dizziness (Nervous system disorders) | 3 (4) | 7 (11)
Cerebrovascular Insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Demyelination (Nervous system disorders) | 1 (1) | 0 (0)
Formication (Nervous system disorders) | 1 (1) | 0 (0)
Hypertensive Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 1 (1)
Intercostal Neuralgia (Nervous system disorders) | 1 (2) | 0 (0)
Migraine (Nervous system disorders) | 1 (4) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 3 (5)
Paraesthesia (Nervous system disorders) | 1 (2) | 4 (4)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Sinus Headache (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar Insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Burning Sensation (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral Atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral Ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Loss Of Consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Tension Headache (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Neurosis (Psychiatric disorders) | 0 (0) | 2 (2)
Panic Attack (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (2) | 0 (0)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast Mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menopausal Symptoms (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Oligomenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Ovarian Cyst Torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal Discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Vaginal Inflammation (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 9 (9)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (6)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal Cord Thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 7 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Dyshidrotic Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pityriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 5 (6)
Pruritus Allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pustular Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 (10) | 0 (0)
Rash Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
Skin Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lichenoid Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pityriasis Rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Swelling Face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tooth Extraction (Surgical and medical procedures) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 8 (8) | 10 (11)
Aortic Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Blood Pressure Fluctuation (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (3) | 1 (1)
Hot Flush (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Raynaud'S Phenomenon (Vascular disorders) | 0 (0) | 1 (1)
Varicose Vein (Vascular disorders) | 0 (0) | 1 (1)
Venous Insufficiency (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least sixty (60) days prior to submitting or presenting a manuscript or other materials relating to the Study to a publisher, reviewer, or other outside persons, the Site shall provide to Sponsor a copy of all such manuscripts and materials, and allow Sponsor sixty (60) days to review and comment on them. If the Sponsor requests, the Site shall remove any Confidential Information (other than Study results) prior to submitting or presenting the materials.